CLINICAL TRIAL: NCT05065242
Title: Smartphone-delivered CBT for Insomnia, a Randomised Controlled Trial
Brief Title: Smartphone-delivered CBT-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Rikard Sunnhed, Lecturer, Adjunct, Psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBT-I - L2S
Record Dates: First submitted 2021-09-09; First posted 2021-10-04 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Cognitive behaviour therapy; Moderation; Mediation; Efficacy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Negotiating | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental): Cognitive Behavior Therapy involves the use of stimulus control and sleep restriction in order to reverse maladaptive sleep habits (time in bed, napping, bedtime variability, rise time variability) proposed to maintain insomnia. It also involves the practice of sleep hygiene principles and to a lesser extent some cognitive exercises. focused on handling sleep disturbing thought activities.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Waitlist (No Intervention): The waitlist serves as a passive control which will receive the same measures as the cognitive behaviour therapy group.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Sleep restriction, Stimulus control, sleep hygiene and cognitive techniques to handle sleep disturbing thoughts.
  Arms: Cognitive Behavioural Therapy

SUMMARY:
The overall purpose with this investigation was to increase access to cognitive behavioural therapy for insomnia (CBT-I) by examining CBT-I delivered through a smartphone application

The first aim that will be addressed is to explore the efficacy of the smartphone delivered CBT-I on overall insomnia and on nighttime symptoms by comparing CBT-I to a waitlist control in a randomised controlled trial.

The second aim is to investigate the effect smartphone delivered CBT-I compared to the waitlist on secondary outcomes related to insomnia, such as stress, anxiety, depression, quality of life and functional impairment.

The third aim that will be addressed is to examine what patient characteristics that CBT delivered to a smartphone depend on to be effective with a treatment-moderator strategy. To investigate moderators, the following moderators will be assessed; age, gender, occupational status, level of education, initial insomnia severity, dysfunction, medication use, chronic pain, somatic/psychiatric co-morbidity, and proposed behavioral mediators of sleep restriction and stimulus control will also be employed as moderators.

The fourth aim that will be addressed is to examine behavioural processes of sleep restriction and stimulus control as potential mediators of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of insomnia more than three nights per week and for more than three months.
* Insomnia despite adequate opportunity to sleep.
* Insomnia severity typical for insomnia disorder, i.e. 11 points or more on the Insomnia Severity Index (ISI).
* Nighttime insomnia symptoms, i.e., two points or more on at least one of the first three ISI questions.
* Daytime insomnia symptoms, i.e. two points or more on one or both of the ISI distress and impairment items (numbers 5 and 7).
* Clinical insomnia symptoms from sleep diaries concerning three nighttime symptoms (difficulties with sleep initiation, difficulties with sleep maintenance, and early morning awakenings), i.e., thirty minutes or more on average on one or more of the symptoms.
* No current or past CBT-I treatment within the past 5 years.
* Time and opportunity to participate in treatment for six weeks.
* Time and opportunity to engage with the treatment content and execute homework assignments for six weeks.
* Access to a smart mobil telephone, email and internet.

Exclusion Criteria:

* Severe depression, i.e., more than 30 points on MADRS-S.
* Suicidal risk, i.e., 4 points or more on item 9 on MADRS-S.
* A high intake of alcohol or caffeine,
* Insomnia due to shiftwork or other sleep-disturbing events (e.g., pregnancy, small children, or animals in the sleep environment).
* Participants with a history of psychotic or bipolar disorder.
* If a somatic condition is reported, it is required that it is relatively stable and/or that the candidate is receiving treatment for the condition.
* When a candidate fulfills criteria for a psychiatric or somatic condition, it is required that insomnia is the disorder currently most distressing and disabling or that the insomnia remains despite treatment for the comorbid condition.
* Participants with the following primary sleep disorders will be excluded via the Duke Structured Interview for Sleep Disorders (DSISD): sleep apnea, restless legs syndrome, periodic limb movement disorder, circadian rhythm disorder, and parasomnias.
* If sleep medication is used, it is required that the use has been relatively stable during three months.
* If Selective Serotonin Reuptake Inhibitors (SSRI) use is reported, it is required that the onset of the medication was at least three months prior to the telephone interview.
* Participants who regularly consume sleep-disturbing medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Insomnia severity index | Pretreatment (week 0), during treatment (i.e., weekly: 1, 2, 3, 4, 5), post-treatment (week 6) and follow-up at 3 month after treatment.
  Global measure of insomnia severity, used for assessing change in insomnia severity from pretreatment to posttreatment.

SECONDARY OUTCOMES:
Work and Social Adjustment Scale | Pretreatment (week 0), post-treatment (week 6) and follow-up at 3 month after treatment
  Score: 0-40, with higher scores indicating worse outcome.
Sleep onset latency (SOL) | Pretreatment (week 0), during treatment (i.e., weekly: 1, 2, 3, 4, 5), post-treatment (week 6).
Wake time after sleep onset (WASO). | Pretreatment (week 0), post-treatment (week 6).
Early morning awakenings (EMA). | Pretreatment (week 0), post-treatment (week 6).
Total sleep time (TST). | Pretreatment (week 0), post-treatment (week 6).
Depression, anxiety and stress scale-21 | Pretreatment (week 0), post-treatment (week 6) and follow-up at 3 month after treatment.
  Score: 0-63, with higher scores indicating worse outcome.
Brunnsviken Brief Quality of life index | Pretreatment (week 0), post-treatment (week 6) and follow-up at 3 month after treatment.
  Score: 0-96, with higher scores indicating better quality of life.
Bed and rise time variability | Pretreatment (week 0), during treatment (i.e., weekly: 1, 2, 3, 4, 5), post-treatment (week 6).
Time in bed (TIB) | Pretreatment (week 0), during treatment (i.e., weekly: 1, 2, 3, 4, 5), post-treatment (week 6).
Pre sleep arousal scale | Pretreatment (week 0), during treatment (i.e., weekly: 1, 2, 3, 4, 5), post-treatment (week 6) and follow-up at 3 month after treatment.
  Score: 16-80, with higher scores indicating worse outcome.

OTHER OUTCOMES:
Credibility Expectancy Questionnaire. | During the first treatment module (first week of treatment).
  Score: 4 items, 1-9, 2 items 0-10, with higher scores indicating higher credibility and expectancy.
Client Satisfaction Questionnaire. | Post-treatment (week 6)
  Score: 8-32, with higher scores indicating higher satisfaction.
Activity and adherence with treatment protocol (self developed questionnaire assessing treatment activity and adherence relating to text, homework and therapist support). | Post-treatment (week 6)
  Score ranging from 1-5, with higher scores indicating higher activity and adherence.
three items assessing sick-leave and other concomitant treatment (self developed questionns). | Post-treatment (week 6) and at 3-month follow-up.
  Item one assessing number of days on sick-leave. Item two assessing whether participants have sought other healthcare options. Item three assessing whether participants have received other treatments for their sleeping issues during the specified time frames.
Adverse events (questionnaire from a previous similar study). | Post-treatment (week 6)
Changes in suicide risk (Item 9 from the MADRS). | Pretreatment (week 0), post-treatment (week 10) and follow-up at 6 month after treatment.
  Score: 0-6, with higher scores indicating a higher suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Sunnhed, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institute, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided